CLINICAL TRIAL: NCT04604054
Title: Comparative Study Between Granulocyte Colony Stimulating Factor and Human Chorionic Gonadotropin in Patients With History of Recurrent Implantation Failure in Intra Cytoplasmic Sperm Injection (at Ovum Pick up Day)
Brief Title: The Effect of Granulocyte Colony Stimulating Factor Versus Human Chorionic Gonadotropin in Females With a History of RIF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Elsayed Eldesouky, Assistant professor of obstetrics and gynecology faculty of medicine Alazhar university Cairo, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 000000415
Record Dates: First submitted 2020-10-22; First posted 2020-10-27 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Fertility Disorders
MeSH Terms: interventions — Chorionic Gonadotropin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Females With a History of Recurrent Implantation Failure in Intra Cytoplasmic Sperm Injection will receive Granulocyte Colony Stimulating Factor as a treatment.
  Interventions: Drug: Granulocyte Colony Stimulated Factor
- Group 2 (Active Comparator): Females With a History of Recurrent Implantation Failure in Intra Cytoplasmic Sperm Injection will receive Human Chorionic Gonadotropin as a treatment.
  Interventions: Drug: Human Chorionic Gonadotropins

INTERVENTIONS:
Drug: Granulocyte Colony Stimulated Factor — GCSF was intrauterine injected once at ovum pick up day
  Other Names: GCSF
  Arms: Group 1
Drug: Human Chorionic Gonadotropins — 500 IU of HCG was injected intrauterine once at ovum pick up day
  Other Names: HCG
  Arms: Group 2

SUMMARY:
One hundred patients who suffered from recurrent implantation failure in intracytoplasmic sperm injection (ICSI) were allocated in the study. On ovum pick-up day, 50 of them were intrauterine injected with granulocyte colony-stimulating factor (G-CSF) and the other 50 were injected with intrauterine Human Chorionic Gonadotropins (HCG). The clinical pregnancy rate was evaluated as a primary outcome and ultrasound imaging of the gestational sac was evaluated as a secondary outcome

DETAILED DESCRIPTION:
One hundred patients suffering from recurrent implantation failure in intracytoplasmic sperm injection (ICSI) were included in the study. The patients were randomly allocated into two groups. The intervention group consisted of 50 patients who received intrauterine injected with granulocyte colony-stimulating factor (G-CSF). The other group (the control group) consisted of 50 patients and injected with intrauterine Human Chorionic Gonadotropins (HCG). Both groups received the interventions at ovum pick-up day. The main outcome was the clinical pregnancy rate which has been evaluated after 2 weeks of the positive pregnancy test. The secondary outcome was an ultrasound image of the gestational sac after 6 weeks of pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Females suffering from recurrent implantation failure and undergoing ICSI

Exclusion Criteria:

* presence of comorbidity as diabetes, hypertension, heart diseases, or endocrine disorders

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-10-30 (Estimated); Primary Completion 2021-01-10 (Estimated); Study Completion 2021-01-10 (Estimated)

PRIMARY OUTCOMES:
clinical pregnancy rate | after 14 days from positive pregnancy test
  number of pregnancies that is confirmed by both high levels of hCG (the pregnancy hormone) and ultrasound confirmation of a gestational sac or heartbeat (fetal pole)

SECONDARY OUTCOMES:
ultrasound image of Gestational sac | 6 weeks of pregnancy
  The gestational sac (GS) is the first sign of early pregnancy on ultrasound